CLINICAL TRIAL: NCT02593708
Title: Phase I Study to Evaluate the Safety of Neratinib in Combination With Paclitaxel, Trastuzumab and Pertuzumab in Women and Men With Advanced or Metastatic HER2+ Solid Tumors
Brief Title: Phase1 of Neratinib+Trastuzumab, Pertuzumab, Paclitaxel in Patients With Advanced Solid Tumors/HER2+
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: toxicity
Sponsor: Michelle Melisko (Other)
Responsible Party: Sponsor-Investigator, Michelle Melisko, Associate Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 149517
Record Dates: First submitted 2015-10-30; First posted 2015-11-02 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Solid Tumor
Keywords: HER2+
MeSH Terms: interventions — neratinib; Paclitaxel; pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cohort 0 (Experimental): 1. Neratinib: 80 mg, daily, oral
  2. Paclitaxel: 80 mg/m2, weekly, intravenously
  3. Pertuzumab: 840 mg loading dose, 420 mg every 3 weeks, intravenously
  4. Trastuzumab: 4 mg/kg loading dose, 2mg/kg every week, intravenously
  Interventions: Drug: Neratinib; Drug: Paclitaxel; Drug: Pertuzumab; Drug: Trastuzumab
- Cohort 1 (Experimental): 1. Neratinib: 120 mg, daily, oral
  2. Paclitaxel: 80 mg/m2, weekly, intravenously
  3. Pertuzumab: 840 mg loading dose, 420 mg every 3 weeks, intravenously
  4. Trastuzumab: 4 mg/kg loading dose, 2mg/kg every week, intravenously
  Interventions: Drug: Neratinib; Drug: Paclitaxel; Drug: Pertuzumab; Drug: Trastuzumab
- Cohort 2 (Experimental): 1. Neratinib: 160 mg, daily, oral
  2. Paclitaxel: 80 mg/m2, weekly, intravenously
  3. Pertuzumab: 840 mg loading dose, 420 mg every 3 weeks, intravenously
  4. Trastuzumab: 4 mg/kg loading dose, 2mg/kg every week, intravenously
  Interventions: Drug: Neratinib; Drug: Paclitaxel; Drug: Pertuzumab; Drug: Trastuzumab
- Cohort 3 (Experimental): 1. Neratinib: 200 mg, daily, oral
  2. Paclitaxel: 80 mg/m2, weekly, intravenously
  3. Pertuzumab: 840 mg loading dose, 420 mg every 3 weeks, intravenously
  4. Trastuzumab: 4 mg/kg loading dose, 2mg/kg every week, intravenously
  Interventions: Drug: Neratinib; Drug: Paclitaxel; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Drug: Neratinib
Drug: Paclitaxel
Drug: Pertuzumab
Drug: Trastuzumab

SUMMARY:
Open label, non-randomized, dose escalation and expansion Phase Ia/b trial to evaluate the safety and tolerability of the combination of neratinib plus paclitaxel, trastuzumab and pertuzumab to determine the recommended Phase II/III dose of this combination.

Neratinib will be given once daily days 1-21 and should be taken orally with food. Paclitaxel and trastuzumab will be given IV on days 1, 8, and 15 out of 21 day cycles. Pertuzumab will be given IV every 3 weeks on day 1 out of 21-day cycles. Each cycle will be 21 days in duration.

Patients will continue on treatment until disease progression or intolerable toxicity.

DETAILED DESCRIPTION:
Neratinib is a potent, irreversible, small molecule panErbB inhibitor of EGFR, HER2 and HER4 tyrosine kinases. Its activity prevents the autophosphorylation of HER2 and thus halts the downstream activation of this key proliferative pathway in tumors dependent on HER2 overexpression or EGFR activation. It has shown promising clinical activity in women with HER2+ stage 2 and 3 breast cancer in the neoadjuvant setting (I-SPY 2 TRIAL) and in women with stage 4 metastatic breast cancer, although evaluation in larger phase 3 trials is required to confirm these results.

The rationale for this study is to determine the feasibility of adding neratinib to a taxane based chemotherapy and the approved HER2 antagonists, trastuzumab and pertuzumab.

The study will evaluate the safety and tolerability and recommended dose of daily neratinib in combination with weekly paclitaxel, trastuzumab and tri-weekly pertuzumab in patients with HER2+ advanced or metastatic disease and, if successful, determine an optimal dose to move into phase II/III testing of this combination in the neoadjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* Women and men 18 years or older with advanced solid tumor malignancy
* Ability to understand and voluntarily sign informed consent prior to undergoing any study-related assessments or procedures, as well as adhere to the study visit schedule and other protocol requirements.
* Local histologic or cytologic confirmation of HER2+ solid tumors by FISH amplification or IHC (3+)
* Patients must have received one prior approved therapy for metastatic disease and have not curable options
* For escalation: Documentation by established staging studies or clinical examination to have measurable or non-measurable metastatic disease per RECIST v1.1 criteria.
* For expansion: Documentation by established staging studies or clinical examination to have measurable metastatic disease per RECIST v1.1 criteria.
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Adequate organ function:
* Absolute neutrophil count (ANC) ≥ 1.5 X 109/L
* Hemoglobin (Hgb) ≥9g/dL
* Platelets (plt) ≥ 100 x 109/L
* Potassium within normal range, or correctable with supplements;
* Serum calcium and magnesium within the normal range (or corrected with supplements)
* AST and ALT ≤2.5 x Upper Limit Normal (ULN)
* Serum total bilirubin ≤ 1.5 x ULN
* Serum creatinine ≤ 1.5 x ULN, or 24-hr clearance ≥ 60ml/min
* Serum albumin > 3.0 g/dL
* Left ventricular ejection fraction of >55% (or institutional lower normal value)
* Females of child-bearing potential (FCBP) must have negative serum pregnancy test within 7 days before starting study treatment and willingness to adhere to acceptable forms or birth control (a physician- approved contraceptive method: oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner)

FCBP is defined as a sexually mature women who:

* Have not undergone a hysterectomy (the surgical removal of the uterus) or bilateral oophorectomy (the surgical removal of both ovaries) or,
* Have not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time during the preceding 12 consecutive months
* Must be willing to practice abstinence or use highly effective contraception for a minimum of 6 months following completion of study treatment (in addition to during study therapy)
* Male subjects with female partner of childbearing potential must agree to the use of a physician-approved contraceptive method throughout the course of the study and for 3 months after the last dose of the investigational product.
* Ability to take oral medications

Exclusion Criteria:

* Any significant medical condition, laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
* Any condition that confounds the ability to interpret data from the study.
* Patients must have recovered from side effects from prior cancer-directed therapy to grade 1 or less (unless deemed not clinically significant by study investigator).
* Symptomatic central nervous system metastases. Subjects with brain metastases that have been previously treated and are stable for 4 weeks are allowed.
* Persistent diarrhea or malabsorption ≥ NCI CTCAE grade 1, despite medical management, ulcerative colitis, inflammatory bowel disease, resection of the stomach or small bowel, or other disease or condition significantly affecting gastrointestinal function.
* Unstable angina, significant cardiac arrhythmia, or New York Heart Association (NYHA) class III or IV congestive heart failure.
* Grade 2 or higher neuropathy
* Known history of: cardiac disease, heart failure or decreased left ventricular ejection fraction, significant clinical arrhythmias
* Prior systemic cancer-directed treatments or investigational modalities ≤ 5 half lives or 4 weeks, whichever is shorter, prior to starting study drug or who have not recovered from grade 2 or higher side effects of such therapy (except alopecia).
* Major surgery ≤ 2 weeks prior to starting a study drug or who have not recovered from side effects of such therapy.
* Known allergic reaction to neratinib, pertuzumab, trastuzumab, paclitaxel, or any of their components.
* Women who are pregnant or breast-feeding.
* Known active Human Immunodeficiency Virus (HIV) infection, Hepatitis B or C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2015-11-03 (Actual); Primary Completion 2017-01-05 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Up to 2 years
  CTCAE v.4.0
Maximum Tolerated Dose | Up to 2 years
  CTCAE v.4.0

SECONDARY OUTCOMES:
Response Rate | Up to 2 years
  RECIST v.1.1

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California, United States